CLINICAL TRIAL: NCT04391959
Title: A Multicenter, Vehicle-controlled, Randomized Study to Evaluate the Safety, Tolerability and Pharmacodynamics of AZR-MD-001 in Patients With Meibomian Gland Dysfunction (MGD)
Brief Title: Evaluation of AZR-MD-001 in Patients With Meibomian Gland Dysfunction (MGD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AZ202001
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2021-01

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZR-MD-001 Vehicle (Experimental): AZR-MD-001 Vehicle will be dosed up to twice weekly.
  Interventions: Drug: AZR-MD-001 Vehicle
- AZR-MD-001 Active (Experimental): AZR-MD-001 Active will be dosed up to twice weekly.
  Interventions: Drug: AZR-MD-001 Active

INTERVENTIONS:
Drug: AZR-MD-001 Active — AZR-MD-001 is an active ophthalmic ointment
  Other Names: AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 Active
Drug: AZR-MD-001 Vehicle — AZR-MD-001 is a vehicle ophthalmic ointment
  Other Names: AZR-MD-001 Vehicle is an ophthalmic ointment
  Arms: AZR-MD-001 Vehicle

SUMMARY:
AZ202001 is a multicenter study of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD)

DETAILED DESCRIPTION:
AZ202001 is a multicenter, double-masked, vehicle-controlled, randomized, parallel group study evaluating the safety, efficacy and tolerability of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Best-corrected visual acuity (BCVA) of 20/40 or better (Snellen equivalent), using the logarithm of the minimum angle of resolution (LogMAR) in each eye
* Evidence of meibomian gland obstruction
* Reported dry eye signs and symptoms within the past 3 months

Exclusion Criteria:

* Uncontrolled ocular disease (except for MGD and dry eye disease/keratoconjunctivitis sicca) or uncontrolled systemic disease
* Glaucoma, ocular hypertension, or intraocular pressure (IOP) in either eye at screening ≥24 mm Hg or has planned insertion/removal of glaucoma filtration shunts/devices during the study
* Corneal abnormality or disorder that impacts normal spreading of the tear film or corneal integrity
* BCVA worse than 20/40 in either eye
* Current use of punctal plugs, anticipated insertion during the study, or a history of punctal cautery in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Tan-Showyin, Principal Investigator — School of Optometry and Vision Science, University of New South Wales
Locations (5):
- Australia (3):
  - Fiona Stapleton, Sydney, New South Wales
  - Scott A Read, Brisbane, Queensland
  - Susan Thackwray, Maroochydore, Queensland
- New Zealand (2):
  - Jagrut Lallu, Auckland
  - Jennifer P Craig, Auckland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active
Started | 16 | 15 (One subject should have been excluded based upon Schirmer test = 0 mm at baseline < 5mm. Subject was removed from the study.)
Completed | 15 | 10
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (13.21) | 56 (20.74) | 57.3 (16.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 9 | 21
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 11 | 9 | 20
  New Zealand | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Meibum Gland Secretion Score (MGS)
Description: Change from Baseline in MGS. The MGS can range from 0 (highly abnormal) to 45 (Normal). Meibomian gland assessment was completed using a handheld instrument, Meibomian Gland Evaluator, along the eyelid margin to ensure measurement consistency. A total of 15 glands will be evaluated along the lower eyelid margin, consisting of 5 glands located in each of the temporal, central and nasal regions, as shown below. For each of the 15 glands, expressed secretion characteristics will be graded on a 0-3 scale. For more detail see: Lane SS, DuBiner HB, Epstein RJ, et al. A new system, the LipiFlow, for the treatment of meibomian gland dysfunction (MGD). Cornea. 2012; 31(4): 396-404.
Time Frame: Month 3
Population: Target Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active
Number analyzed (Participants) | 3 | 4
score on a scale | 0.5 (1.83) | 7.4 (1.53)

2. Secondary Outcome: Total OSDI
Description: Change from Baseline in Total Ocular Surface Disease Index (OSDI). The Total OSDI can range from 0 (normal) to 100 (abnormal). The OSDI questionnaire consists of 12 questions regarding ocular symptoms, environmental triggers, and vision-related functioning. The patient was asked to rate each symptom using a 5-point scale (0 to 4), where 0 = none of the time; 1 = some of the time; 2 = half of the time; 3 = most of the time; and 4 = all of the time. Seven questions related to visual functioning allow a response of "N/A" (not applicable). The total OSDI was calculated from the raw scores of each of the 12 questions based on the formula: ([sum of scores for all questions answereda] X 100)/([total number of questions answered] X 4).
  Questions answered with N/A were excluded in the calculation of total OSDI.
Time Frame: Day 14 to Month 3
Population: Target Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active
Number analyzed (Participants) | 3 | 4
score on a scale | -2.0 (3.49) | -8.1 (2.86)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15
Other Adverse Events (participants affected / at risk) | 2/16 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZR-MD-001 Vehicle (N=16) | AZR-MD-001 Active (N=15)
dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) — This subject experienced dysuria, severe in severity, which was considered unrelated to either the investigational product or the study procedure. After subject hospitalization for transurethral resection of the prostate, the TEAE resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZR-MD-001 Vehicle (N=16) | AZR-MD-001 Active (N=15)
Eye irritation (Eye disorders) | 1 (1) | 2 (2)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 4 (4)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2)
Foreign body sensation (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04391959/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT04391959/SAP_001.pdf